CLINICAL TRIAL: NCT00141752
Title: Toronto Bedside Swallowing Screening Test (TOR-BSST) - A Bedside Swallowing Screening for Stroke Patients
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Stroke Network (Other); Toronto Rehabilitation Institute (Other); Parkwood Hospital, London, Ontario (Other); Sunnybrook Health Sciences Centre (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: CSN II.10
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2012-01

CONDITIONS: Cerebrovascular Accident; Deglutition Disorders
Keywords: Cerebrovascular Accident; Deglutition Disorders; stroke; dysphagia; screening
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Toronto Bedside Swallowing Screening Test (TOR-BSST) — Toronto Bedside Swallowing Screening Test

SUMMARY:
This research will assess the accuracy of the Toronto Bedside Swallowing Screening Test (TOR-BSST), a new dysphagia screening test for patients with stroke. The purpose of the TOR-BSST is to predict the presence of dysphagia in stroke patients across their continuum of care in a simple and efficient manner. This initial research will assess the accuracy of the TOR-BSST in the acute and rehabilitative settings using videofluoroscopy as the gold standard for comparison. The results from this research will also assess the stability of the TOR-BSST across nursing, its primary user, and generate an estimate for the prevalence of dysphagia in adult stroke patients in the acute and rehabilitative settings. Participants in this research will be 315 stroke patients from several teaching centres in Ontario, namely 105 acute patients from the University Health Network, Sunnybrook & Women's College Health Sciences Centre, and Hamilton General Hospital, and 210 patients in the rehabilitation setting from the Toronto Rehabilitation Institute and Parkwood Hospital, London. Both the TOR-BSST and videofluoroscopic assessment will be administered within 24 hours of each other and interpreted according to published preferred practice guidelines for dysphagia. This research will be the first to implement and assess a standardised method for screening for dysphagia in stroke patients across the continuum of stroke recovery.

ELIGIBILITY:
Inclusion Criteria:

* patients with a new diagnosis of brainstem or cerebellar stroke
* patients with a new diagnosis of cortical stroke with NIH Stroke Scale score of 4 or above

Exclusion Criteria:

* patients with a previous history of stroke with dysphagia
* patients with a confirmed history of Parkinson's, Parkinsonian Syndrome, ALS, MSA, MS, dementia, or other neurodegenerative disease
* patients with a history of cranial neurosurgery
* patients with a known previous or current oropharyngeal dysphagia due to structural or neurological cause
* patients with active COPD or current pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly admitted patients with a diagnosis of stroke (refer to eligibility criteria)
Sampling Method: Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2002-10; Primary Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Martino, PhD, Principal Investigator — University of Toronto; Nicholas E Diamant, MD, Principal Investigator — University Health Network, Toronto
Locations (5):
- Canada (5):
  - Hamilton General Hospital, Hamilton, Ontario
  - Parkwood Hospital, London, Ontario
  - Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario
  - Toronto Rehabilitation Institute, Toronto, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario

REFERENCES:
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Martino R, Pron G, Diamant N. Screening for oropharyngeal dysphagia in stroke: insufficient evidence for guidelines. Dysphagia. 2000 Winter;15(1):19-30. doi: 10.1007/s004559910006. PMID 10594255